CLINICAL TRIAL: NCT07207252
Title: Sleep & Stress Test
Brief Title: Research on Sleep and Emotion Testing of Tea Theanine Casein Hydrolysate Pressed Candy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Collaborators: Nu Skin Enterprises (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W24002001
Record Dates: First submitted 2025-09-16; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mild to Moderate Sleep Disorder; Pressure
Keywords: Tea Theanine; Casein Hydrolysate; EEG; Emotion; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tea Theanine Casein Hydrolysate Pressed Candy (Experimental): Take 4 Tea Theanine Casein Hydrolysate Pressed Candies once a day.
  Interventions: Dietary Supplement: Tea Theanine Casein Hydrolysate Pressed Candy
- Pressed Candy (Placebo Comparator): Take 4 Pressed Candies once a day.
  Interventions: Dietary Supplement: Pressed Candy

INTERVENTIONS:
Dietary Supplement: Tea Theanine Casein Hydrolysate Pressed Candy — Take 4 candies once a day. It is recommended to consume it one hour before bedtime.
  Arms: Tea Theanine Casein Hydrolysate Pressed Candy
Dietary Supplement: Pressed Candy — Take 4 candies once a day.
  Arms: Pressed Candy

SUMMARY:
The study evaluates the improvement of sleep, emotion, and skin by standardizing the use of the blend (Tea Theanine Casein Hydrolysate Pressed Candy, whose active ingredients include Tea Theanine, Casein Hydrolysate, and Saffron Extract).

This is a randomized, double-blind trial for Chinese people aged 20-55. The change of sleep, emotion, skin, and other related indicators of 90 participants after taking Tea Theanine Casein Hydrolysate Pressed Candy, whose active ingredients include tea theanine, casein hydrolysate, and saffron extract, was evaluated through a 28 days product placement test (sub study 1), and the emotional change of 70 participants after taking Tea Theanine Casein Hydrolysate Pressed Candy was evaluated through an EEG test (sub study 2).

Participants who meet the inclusion criteria were randomly assigned to use the experimental product or the placebo control. In sub study 1, 90 participants completed a 7-day baseline period, a 28-day testing period (T1d, T7d, and T28d). In sub study 2, 71 participants completed a single on-site test.

ELIGIBILITY:
Sub study 1:

Inclusion Criteria:

1. Chinese participants aged 20-55,
2. Mild to moderate sleep disorders (Pittsburgh Sleep Quality Index 5-21),
3. At least 2/3 of the population is under pressure (PSS-10 ≥ 14),
4. No plans to leave Shanghai in the past three months,
5. Have basic Chinese reading comprehension and expression abilities and can independently complete the questionnaire survey,
6. Voluntarily participate in the test and sign an informed consent form,
7. Willing to comply with all evaluation requirements, use the product according to the research protocol, and complete testing and follow-up. During the trial period, do not change the original dietary or skincare habits or use other similar foods, health products, or drugs.

Exclusion Criteria:

1. Have used any food, health products, or medication with sleep aid and emotional relief effects within one month before the test,
2. History of tea allergy,
3. History of dairy product allergies,
4. Due to occupational reasons requiring night work or regular changes in working hours,
5. Regularly staying up late within one month before the test (not due to objective reasons or negative emotions, the frequency of staying up late is greater than once per week, such as playing games, watching TV shows, etc.),
6. Intending to become pregnant, or currently pregnant or breastfeeding,
7. Currently treating diseases other than sleep disorders,
8. Using facial and eye skincare products with whitening and spot-removing effects,
9. Has a history of alcohol abuse,
10. There were unhealed skin lesions on the face currently,
11. Have undergone surgical procedures, plastic surgery, or organ transplantation in the past year,
12. Any other health problems or chronic illnesses other than sleep and emotions,
13. Other iatrogenic reasons considered by the expert or professional may influence the evaluation outcome.

Sub study 2：

Inclusion Criteria:

1. Chinese participants aged 23-55,
2. Right-handedness (not acquired through training),
3. Pressure group (PSS-10 ≥ 14),
4. No plans to leave Shanghai in the past three months,
5. Have basic Chinese reading comprehension and expression abilities, and can independently complete the questionnaire survey,
6. Voluntarily participate in the test and sign an informed consent form,
7. Willing to comply with all evaluation requirements, use the product according to the research protocol, and complete testing.

Exclusion Criteria:

1. Have used any food, health products, or medication with sleep aid and emotional relief effects within one month before the test,
2. History of tea allergy,
3. History of dairy product allergies,
4. Unable to effectively induce negative emotions during on-site testing (POMS stress scale and panic scale scores after emotional induction are not higher than baseline),
5. Before testing, any obvious physiological discomfort, including but not limited to fever, hunger, dysmenorrhea, cough, lack of sleep, etc.,
6. Frequent insomnia and irregular sleep patterns within a month,
7. Anemia,
8. Abnormal blood sugar and blood pressure,
9. Neurological disorders,
10. Self-reported neurological or emotional disorders such as depression, anxiety, bipolar disorder, and obsessive-compulsive disorder diagnosed by clinical psychiatrists,
11. Alcohol, cigarette addiction, or drug dependence,
12. During drug treatment, ①The individual has systematically taken hypnotic drugs (barbiturates, etc.) or other central nervous system drugs within one year. ②The individual has systematically used anti-anxiety drugs (Benzodiazepines such as diazepam, chlorpromazine, and clonazepam), antiepileptic drugs (such as phenobarbital or clonazepam), antipsychotic, antidepressant, and anti-dementia drugs within one year.
13. Intending to become pregnant, or currently pregnant or breastfeeding,
14. Other iatrogenic reasons considered by the expert or professional may influence the outcome of the evaluation.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Change in scores of Pittsburgh Sleep Quality Index, PSQI (28 Days Product Placement Test) | T0 (baseline before consumption), T1wk (after consumption for 1 week), T4wk (after consumption for 4 weeks)
  The total score range is 0-21 points. The higher the score, the worse the sleep quality.
Change in scores of Restorative Sleep Questionnaire Weekly Version (RSQ-W) and Daily Version (RSQ-D) (28 Days Product Placement Test) | T0 (baseline before consumption, RSQ-W was used), T1d (after consumption for one day, RSQ-D was used), T1wk (after consumption for one week, RSQ-W was used), T4wk (after consumption for four weeks, RSQ-W was used)
  The total score is calculated based on the average score of the questionnaire items, and then the average score is converted to a 0-100 scale using the formula: (average score - 1) * 25. The total score ranges from 0 to 100, with higher scores indicating better restorative sleep.
Change in the Fall asleep time, Nighttime sleep duration, Shallow sleep duration, Shallow sleep ratio and Sleep latency (28 Days Product Placement Test) | Continuous collection during placement (7-day baseline+28-day product placement test)
  These indicators were collected by Huawei Smart Band HA580.
Change in the Wakefulness frequency, Sleep quality, Sleepiness in the morning, Refreshment in the morning, mood in the morning, Sleep latency (28 Days Product Placement Test) | Continuous collection during placement (7-day baseline+28-day product placement test)
  The sleep status of participants was tracked through sleep diaries.
Change in the scores of Perceived Stress Scale, PSS-10 (28 Days Product Placement Test) | T0 (baseline before consumption), T1wk (after consumption for one week), T4wk (after consumption for four weeks)
  The total score is calculated based on the cumulative score of the questionnaire items, ranging from 0 to 40 points, with higher scores indicating greater perceived stress.
Change in the scores of The State-Trait Anxiety Inventory, the S-Form, S-AI (28 Days Product Placement Test) | T0 (baseline before consumption), T1d (after consumption for one day), T1wk (after consumption for one week), T4wk (after consumption for four weeks)
  The total score is calculated based on the cumulative score of the questionnaire items, ranging from 20 to 80 points, with higher scores indicating greater anxiety.
Change in the scores of Profile of Mood States, POMS (28 Days Product Placement Test) | T0 (baseline before consumption), T1d (after consumption for one day), T1wk (after consumption for one week), T4wk (after consumption for four weeks)
  The total score is calculated based on the cumulative score of the questionnaire items, ranging from 56 to 216 points. Higher scores indicate stronger negative emotions, reflecting a depressed mood and feelings of irritability.
Change in the Skin tone evenness, Glossiness, ITA°, L, a, b, Dark circles (Under orbital pigmentation area) ITA°, L (28 Days Product Placement Test) | T0 (baseline before consumption), T1wk (after consumption for 1 week), T4wk (after consumption for 4 weeks)
  All-face skin images under different light sources were captured by VISIA-CR (CANFIELD, America).
Change in the Protrusion volume in Eye bag area (28 Days Product Placement Test) | T0 (baseline before consumption), T1wk (after consumption for 1 week), T4wk (after consumption for 4 weeks)
  Protrusion volume in Eye bag area was measured by Primos (CANFIELD, America).
Change in the Skin smoothness, softness, glossiness, hydration, tone evenness, Overall appearance (28 Days Product Placement Test) | T0 (baseline before consumption), T1wk (after consumption for 1 week), T4wk (after consumption for 4 weeks)
  Dermatologists score the facial skin condition of participants using validated assessment scales (VAS). Scores for each dimension range from 0 to 9, and higher scores reflect a better skin condition.
The improvement of dark circles and eye bags (28 Days Product Placement Test) | T1wk (after consumption for 1 week), T4wk (after consumption for 4 weeks)
  Dermatologists evaluate the improvement of dark circles and eye bags in participants through baseline and follow-up visit VISIA photos, using an integrated visualization system (IVS) with improved investigator visual score. Each score range from 0 to 3, and higher scores represent a higher level of improvement.
Change in the scores of Profile of Mood States, POMS (EEG Test) | Before emotional induction (only tension and confusion scales), immediately after emotional induction, and 60 minutes after using the product
  The sore of tension subscale ranges from 0 to 24 and confusion subscale ranges from 0 to 20, with higher scores indicating greater tension/confusion. The total score is calculated based on the cumulative score of the questionnaire items, ranging from 56 to 216 points. Higher scores indicate stronger negative emotions, reflecting a depressed mood and feelings of irritability.
Change in the Brain wave α power (EEG Test) | During emotion inducting, 60 minutes after consuming the product
  EEG data was collected by Emotiv EPOC X, which is a wireless portable electroencephalograph used for scalable and contextualized brain research, with 14 channels on a 10-20 system, using saline electrode caps and a sampling rate set to 256 SPS. Electrodes were placed according to the electrode positioning of the 10-20 system.
Change in the Brain wave β power (EEG Test) | During emotion inducting, 60 minutes after consuming the product
  EEG data was collected by Emotiv EPOC X, which is a wireless portable electroencephalograph used for scalable and contextualized brain research, with 14 channels on a 10-20 system, using saline electrode caps and a sampling rate set to 256 SPS. Electrodes were placed according to the electrode positioning of the 10-20 system.
Change in the Brain wave θ power (EEG Test) | During emotion inducting, 60 minutes after consuming the product
  EEG data was collected by Emotiv EPOC X, which is a wireless portable electroencephalograph used for scalable and contextualized brain research, with 14 channels on a 10-20 system, using saline electrode caps and a sampling rate set to 256 SPS. Electrodes were placed according to the electrode positioning of the 10-20 system.
Change in the Brain wave θ/β power ratio (EEG Test) | During emotion inducting, 60 minutes after consuming the product
  EEG data was collected by Emotiv EPOC X, which is a wireless portable electroencephalograph used for scalable and contextualized brain research, with 14 channels on a 10-20 system, using saline electrode caps and a sampling rate set to 256 SPS. Electrodes were placed according to the electrode positioning of the 10-20 system.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided